CLINICAL TRIAL: NCT01531907
Title: Relationships Between GLP-2 and Markers of Bone Turnover Following Feeding: the Influence of Obesity and Cellular Mechanisms of Action
Brief Title: Relationships Between GLP-2 and Markers of Bone Turnover Following Feeding
Acronym: GLP-2
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH16160
Record Dates: First submitted 2012-02-03; First posted 2012-02-13 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obesity
Keywords: GLP2; Obesity; Premenopausal; Bone; Formation; Resorption
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — On completion of the study, serum and plasma aliquots will be moved to the Human Tissue Authority (HTA) licensed biorepository housed in the Centre for Biomedical Research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese: Premenopausal women, 25 - 40 years with BMI of ≥30kg/m2
  Interventions: Other: Study visit procedures
- Lean: Premenopausal women, 25 - 40 years with BMI of 18.5-24.9 kg/m2
  Interventions: Other: Study visit procedures

INTERVENTIONS:
Other: Study visit procedures — Anthropometric measurements to include:
  * Weight, height, and BMI.
  * Waist and hip circumference
  * Triceps skinfold thickness
  * Measurement of supine abdominal thickness A baseline blood sample (15ml)is taken before receiving a standard polycal drink (75g glucose load) Three further blood samples (15 ml) will be taken, at the time points 20, 60 and 120 minutes after glucose loading. In 10 subjects (5 lean and 5 obese) we will take an additional blood sample (up to 50 ml) at baseline into heparin to grow osteoclasts in culture. Visit duration - approximately 3-4 hours.

SUMMARY:
This study has been designed to study differences bone turnover in relation to glucagon-like peptide-2 (GLP-2) following feeding in lean and obese premenopausal women. Given the preliminary evidence that GLP-2 may act directly on osteoclasts, the investigators plan to determine whether GLP2 receptors are expressed in osteoclasts and the effect of GLP-2 on bone resorption.

Hypotheses:

1. Acute responses of GLP-2 and bone resorption markers following feeding are affected by body fat mass.
2. Serum levels of GLP-2 are lower in obese pre-menopausal women and are associated with a reduction in trabecular and/or cortical bone mass
3. GLP-2 has direct actions on osteoclast resorption via a functional receptor

DETAILED DESCRIPTION:
Study objectives:

1. To determine if differences in baseline serum levels of GLP-2 are related to differences in bone microarchitecture, structure and strength at the distal tibia and distal radius between obese and lean premenopausal females.
2. To determine whether obesity in premenopausal females influences levels of circulating GLP-2 following a standardised glucose meal with a resultant change in markers of bone formation and resorption
3. To test whether GLP-2 directly affects osteoclast function via an identifiable receptor

ELIGIBILITY:
Inclusion Criteria:

* Age 25-40
* Caucasian
* Premenopausal
* Able and willing to consent
* BMI either 18.5-24.9 kg/m2 or ≥30 kg/m2
* Completion 'The Effects of Obesity on Bone Structure and Strength' study REC ref 10/H1308/61
* Consented to be approached for future research studies

Exclusion Criteria:

* Fracture less than twelve months prior to recruitment
* History of any long term immobilization (duration greater than three months)
* Current pregnancy or trying to conceive Pregnancy or breast feeding less than one year prior to recruitment
* Diabetes mellitus
* History of or current conditions known to affect bone metabolism, which may include:

  * Diagnosed skeletal disease or osteoarthritis
  * Chronic renal disease
  * Acute or chronic hepatic disease
  * Hyperparathyroidism or Hyperthyroidism
  * Malabsorption syndromes
  * Diagnosed endocrine disorders
  * Diagnosed diabetes mellitus
  * Clinically significant hypocalcemia or hypercalcemia
  * Diagnosed restrictive eating disorder
* Current or clinically significant previous use of medications or treatment known to affect bone metabolism, for example:

  * Depot medroxyprogesterone or the combined oral contraceptive pill
  * Glucocorticoid therapy
  * Anti-convulsant therapy
  * Bone treatments (e.g. Bisphosphonates)
* Alcohol intake of greater than 21 units per week
* Athlete, defined as an individual participating in competitive sport at amateur or professional level
* Monogenic and obesity syndromes
* History of cancer within the past 5 years excluding skin cancer non melanomas

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators will recruit healthy pre-menopausal, Caucasian female participants 25-40 years and divide them into two groups, obese and lean according to their Body Mass Index. Participants will be identified and approached from a study group of obese and lean participants previously recruited for the 'The Effects of Obesity on Bone Structure and Strength - Fat and Bone Study (FAB)' study (REC ref 10/H1308/61) conducted at the Academic Unit of Bone Metabolism (AUBM) in Sheffield. Participants from this study have been selected as some of the scan and neuromuscular function data generated from this study will be reused as explained below. Body Mass Index ≥30 kg/m2 will be used to define obesity with BMI for lean participants defined as 18.5-24.9 kg/m2. Thirty participants will be recruited, 15 obese and 15 lean. Participants will be matched for age, and where possible height.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
GLP-2 levels | Change at 20, 60 and 120 minutes

SECONDARY OUTCOMES:
Osteocalcin levels | Change at 20, 60 and 120 minutes
β Carboxy-terminal collagen crosslinks (β CTx)levels | Change at 20, 60 and 120 minutes
Procollagen 1 N-terminal propeptide (P1NP) levels | Change at 20, 60 and 120 minutes
High-resolution peripheral quantitative computed tomography (HRpQCT) | At baseline
Dual-emission X-ray absorptiometry (DXA) | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dimitri, Dr, Principal Investigator — Sheffield Childrens Hospital
Locations (1):
- Academic Unit of Bone Metabolism, Sheffield, South Yorkshire, United Kingdom